CLINICAL TRIAL: NCT01405495
Title: Posttraumatic Stress Disorder (PTSD) Among Victims of Sexual Abuse and Changes in Structural and Functional Brain Connectivity: A Cognitive and Neuroanatomical Markers Study Using fMRI,(DTI) and(ASL)
Brief Title: PTSD Among Victims of Sexual Abuse and Changes in Structural and Functional Brain Connectivity
Acronym: COPTSD
Status: Completed | Type: Observational
Sponsor: University Hospital, Tours (Other)
Responsible Party: Sponsor
Other Study IDs: PHRI/10/WEH/COPTSD
Record Dates: First submitted 2011-06-07; First posted 2011-07-29 (Estimated); Last update posted 2017-05-04 (Actual); Status verified 2017-05

CONDITIONS: PostTraumatic Stress Disorder
Keywords: Posttraumatic Stress Disorder; Working Memory; Attentional Bias; Connectivity; Structural Neuroimaging; Functional Neuroimaging; Diffusion Tensor Imaging; Arterial Spin Labelling; Cortisol; Psychophysiology; Early development of
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Diffusion Tensor Imaging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Salivary cortisol
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- PTSD group: Intervention 'MRI-based techniques (sMRI, fMRI, DTI, ASL)'
  Interventions: Procedure: MRI-based techniques (sMRI, fMRI, DTI, ASL)
- Exposed without PTSD: Intervention 'MRI-based techniques (sMRI, fMRI, DTI, ASL)'
  Interventions: Procedure: MRI-based techniques (sMRI, fMRI, DTI, ASL)
- Healthy Controls: Intervention 'MRI-based techniques (sMRI, fMRI, DTI, ASL)'
  Interventions: Procedure: MRI-based techniques (sMRI, fMRI, DTI, ASL)

INTERVENTIONS:
Procedure: MRI-based techniques (sMRI, fMRI, DTI, ASL) — no drugs include
  Other Names: structural magnetic resonance imaging; functional magnetic resonance imaging; diffusion tensor imaging; arterial spin labelling

SUMMARY:
The goal of this study is to identify the early modifications in fronto-temporal connectivity in female victims who developed PTSD, compared to female victims who did not develop the disorder, and to healthy control females. The investigators will compare between all these groups, structural and functional differences using different techniques (MRI, fMRI, DTI and ASL), and paradigms (cognitive tasks or at rest).

DETAILED DESCRIPTION:
Most of the transversal neuroimaging studies in posttraumatic stress disorder (PTSD) were conducted in male war veterans. Few studies focused on neuroanatomical correlates of PTSD in civilian populations, and only one prospective study explored the cerebral connectivity when developing the disorder. In France, physical and sexual assaults are the most prevalent causes of PTSD, especially in the female population. Neuroanatomic basis of chronic PTSD are now well-defined, implicating limbic over-activation (amygdala), associated with a default activation in prefrontal cortex. However, mechanisms implied in the modification of fronto-limbic regions connectivity, especially in the anterior cingulate cortex (ACC), need further investigations. Will the post-traumatic amygdalar over-activation perturbate the normal functioning of the ACC, or is there a modification in the ACC functioning which leads to a default in amygdala inhibition ? This question is of interest, since the prefrontal cortex, including the ACC, has an essential role in different kind of cognitive activities in the normal and pathological brain, such as working memory and attentional processes.

The goal of this study is to characterize early modifications in structural and functional connectivity in brain structures implied in the development of PTSD using different kinds of MRI-based techniques (structural MRI, fMRI, DTI and ASL), as well as biological (cortisol) and psychophysiological (skin conductance ...) measures in female patients developing PTSD, compared to women exposed to trauma who did not develop the disorder and to healthy controls.

ELIGIBILITY:
Inclusion Criteria:

* Written consent
* affiliated to the National Health Insurance
* without neurological past history
* without psychoactive drugs past history

Exclusion Criteria:

* the subject can not follow the instructions
* simultaneous participation to an other study using psychoactive drugs
* blindness
* epilepsy
* addiction to psychoactive drugs
* MRI counter-indications (pace-makers ...)
* claustrophobia
* every circumstances making the subject unable to understand the nature, the objectives or the consequences of the study

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: PTSD related to sexual abuse vs trauma-exposed vs controls, in right-handed females.
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2012-02; Primary Completion 2016-02 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Changes from baseline brain connectivity in sexual assault female victims who developed PTSD compared to victims without PTSD and healthy control at 6 months. | One month (plus or minus 2 weeks) and 6 months (plus or minus 2 weeks) post trauma
  We will measure differences in cerebral functional (fMRI) and morphologic (DTI) connectivity during cognitive tasks or at rest in the different groups of participants. It will allow us to understand what are the specific connectivity differences induced by the disorder, but also by the exposition to a traumatic event, compared to healthy controls.

SECONDARY OUTCOMES:
Changes from baseline cerebral activity between groups during cognitive tasks and difference between groups in measures of specific brain structure volumes at 6 months. | One month (plus or minus 2 weeks) and 6 months (plus or minus 2 weeks) post trauma
  We will measure differences in cerebral activity during cognitive tasks in the different groups of participants. It will allow us to understand what are the specific differences induced by the disorder, but also by the exposition to a traumatic event, compared to healthy controls. Also, according to the literature, we will measure the differences in specific brain structure volumes (e.g., hippocampus)between the different groups.

CONTACTS AND LOCATIONS:
Overall Officials: Wissam El-Hage, MD, PhD, Principal Investigator — INSERM U930 Team 4 Affective Disorders
Locations (1):
- Bretonneau Regional Universitary Hospital, Tours, France